CLINICAL TRIAL: NCT05562375
Title: Predictive Value of GOCCLES® (Glasses for Oral Cancer Curing Light Exposed Screening), Device for Early Diagnosis of Oral Potentially Malignant Disorders
Brief Title: Predictive Value of GOCCLES® Device for Early Diagnosis of Oral Potentially Malignant Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Rocío Teresa Martín Munoz, Bachelor of Dentistry and Specialist in Oral Medicine, Universidad Rey Juan Carlos
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3011202123121
Record Dates: First submitted 2022-09-22; First posted 2022-09-30 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Oral Potentially Malignant Disorders; Oral Cancer
Keywords: GOCCLES; Autofluorescence; Oral cancer; Oral dysplasia
MeSH Terms: conditions — Mouth Neoplasms | interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): 73 patients are to be recruited from the ones that go to the oral medicine service at the university clinic of Rey Juan Carlos in Madrid that present a compatible clinic diagnostic compatible with oral potentially malignant disorders. Each patient will receive first an intraoral exploration, taking note of location and size of the injury. After that, an exploration with the GOCCLES® device will be made, also taking note of the location and size data. Thereafter, the blue toluidine stain will be used, taking note of the size and location of the marked areas. Pictures will be taken through all the steps. Finally, a biopsy will be made of the area or areas the clinic considers and/or marked by the device or the toluidine blue.
  Interventions: Device: GOCCLES; Diagnostic Test: Toluidine blue stain; Procedure: Biopsy

INTERVENTIONS:
Device: GOCCLES — Inspection using GOCCLES®. An UV light source will be administered, with polymerization lamp sdi radii xpert, with a potency of 1500 mW/cm2 and a wavelength of 440-480nm, applied at 20cm of the injury.
  Notes will be taken on the location and size of the injury observed with the device.
  Image register using the GOCCLES® photographic filter for mobile devices. The same light source will be used.
Diagnostic Test: Toluidine blue stain — To value the toluidine blue diagnosis capacity, the sequence described by Mashberg will be followed: The patient will realize a mouthwash with acetic acid at 1% for 20 seconds. Two using water for 20 seconds. Toluidine blue at 1% will be applied for 20 seconds. New mouthwash with acetic acid for 60 seconds and a final mouthwash with water.
  Notes on the and pictures will be taken on the location and size of the injury.
Procedure: Biopsy — The area to biopsy will be chosen, and, using local anaesthesia, it will be resected. The specimens will be sent to the oral and maxillofacial pathology diagnostic service of the University of Basque Country for anatomopathological study

SUMMARY:
Oral potentially malignant disorders (OPMDs) are chronic pathologies which can suffer dysplastic alterations and evolve into oral cancer.

The diagnosis of those pathologies is commonly done by visual inspection, which is not capable of determining the presence or not of dysplasia. Furthermore, this type of diagnosis depends greatly on the expertise and training of the professional.

In recent years, new methods that can help early oral cancer diagnosis have been developed. A new device has been commercialized, named GOCCLES® (Glasses for Oral Cancer Curing Light Exposed Screening), based on the autofluorescence principle.

The hypothesis of this study is that GOCCLES® device could be an effective tool to help in early detection of oral cancer.

DETAILED DESCRIPTION:
The main objective of this study is to establish GOCCLES® autofluorescence method predictive value in early diagnostic of malignant oral disorders and/or potentially malignant oral cavities.

The secondary objectives are comparing the match in zone detection between this method and blue toluidine staining, and valuing if blue toluidine staining brings additional information to the dysplastic injuries diagnoses when combined to the GOCCLES® device.

This study will follow the STARD (Standards for Reporting of Diagnostic Accuracy Studies) guideline.

It is intended to recruit 73 patients from the oral medicine service at the university clinic of Rey Juan Carlos University in Madrid, that present a compatible clinic diagnostic with oral potentially malignant disorders. Each patient will receive first an intraoral exploration, taking note of location and size of the injury. After that, an exploration with the GOCCLES® device will be made, also taking note of the location and size data. Thereafter, the blue toluidine stain will be used, taking note of the size and location of the marked areas. Pictures will be taken through all the steps. Finally, a biopsy will be made of the area or areas the clinic considers and/or marked by the device or the toluidine blue.

DETAILED PROCEDURE:

1. Specific location of the injury or injuries will be taken.
2. Its maximum size will be measured.
3. Photographic record with Canon EFS 60mm camera and Canon Macro Ring Lite MR-14EX ring flash.
4. Inspection using GOCCLES®. An UV light source will be administered, with Sdi Radii Xpert polymerization lamp with a potency of 1500mW/cm2 and a wavelength of 440-480nm, applied at 20cm of the injury.
5. Notes will be taken on the location and size of the injury observed with the device.
6. Image register using the GOCCLES® photographic filter for mobile devices. The same light source will be used.
7. To value the toluidine blue diagnosis capacity, the sequence described by Mashberg will be followed: The patient will realize a mouthwash with acetic acid at 1% for 20 seconds. Two using water for 20 seconds. Toluidine blue at 1% will be applied for 20 seconds. New mouthwash with acetic acid for 60 seconds and a final mouthwash with water.
8. Notes on the and pictures will be taken on the location and size of the injury.
9. The area to biopsy will be chosen, and, using local anaesthesia, it will be resected.
10. The sample or samples will be sent to the Oral and Maxillofacial Pathology Diagnostic Service of the University of the Basque Country, properly preserved in formalin and with the corresponding report.
11. In addition, the following data of each patient will be registred: age, sex, harmful habits, medical history of interest, type of injury, location of the injury, size of the injury and presumptive diagnosis.

If the area chosen by the investigator as the most adequate one matches the one referred by the GOCCLES® glasses and the toluidine blue, only one biopsy will be made. Otherwise, two or three samples will be taken. The patient will be called after 7-15 days, to receive the results and the retiring of the suture if required, and to start treatment in cases which it is needed.

A lesion will be considered positive if, when using GOCCLES® device, a loss of fluorescence is observed in an area or areas of the lesion, that is, when a brownish, brown or dark brown area or areas are observed.

A lesion will be considered to be positive for toluidine blue staining when, after carrying out the sequence described by Mashberg, an intense blue staining is produced in an area or areas of the lesion

A positive result will be considered after performing biopsy in those cases in which the anatomopathological analysis indicates the presence of dysplasia, whatever its grade, or the presence of malignant transformation.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18.
* Patients that present oral mucosa injuries compatible with OPMD.
* Patients that understand the purpose of the study and express consent

Exclusion Criteria:

* Patients that don't have the capability to express consent.
* Patients with systemic pathologies that contraindicate a biopsy.
* Patients with a recent biopsy at the oral cavity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2022-01-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Intraoral examination. Location of the lesion | This procedure will be realised in the first appointment, at day 1, and it will take a time of five minutes
  Intraoral examination of the injury with white light. Information about location will be recorded in a data collection document, individual for each patient.
Intraoral examination. Size of the lesion | This procedure will be realised in the first appointment, at day 1, and it will take a time of five minutes
  Intraoral examination of the injury with white light. The size of the injury will be measured with an acetate rule. This information will be recorded in a data collection document, individual for each patient.
Intraoral examination. Photographic record | This procedure will be realised in the first appointment, at day 1, and it will take a time of five minutes
  Photographs of the lesion will be recorded with a Canon EFS 60 mm camera and Canon Macro Ring Lite MR-14EX ring flash
Oral examination with GOCCLES device | This procedure will be realised in the first appointment, at day 1, immediately after intraoral examination, and it will take a time of ten minutes.
  An UV light source will be administered, with polymerization lamp sdi radii xpert, with a potency of 1500 mW/cm2 and a wavelength of 440-480nm, applied at 20cm of the injury. Notes will be taken on the location and size of the injury observed with the device.
  Image register using the GOCCLES® photographic filter for mobile devices. The same light source will be used.
Toluidine blue staining of the lesion | This procedure will be realised in the first appointment, at day 1, immediately after oral examination with GOCCLES device, and it will take a time of fifteen minutes.
  For this procedure, Mashberg technique will be realised. The patient will realize a mouthwash with acetic acid at 1% for 20 seconds. Two using water for 20 seconds. Toluidine blue at 1% will be applied for 20 seconds. New mouthwash with acetic acid for 60 seconds and a final mouthwash with water. Information about location and size of the stained area will be recorded in the data collection document. Photographs will be taken with the Canon EFS 60mm camera and Canon Macro Ring Lite MR-14EX ring flash.
Biopsy and histopathological analysis | This procedure will be realised in the first appointment, at day 1, immediately after de toluidine blue staining, and it will take a time of twenty minutes. The patient will be called after 7-15 days, to receive the results.
  The area to biopsy will be chosen, and, using local anaesthesia, it will be resected. If the area chosen by the investigator as the most adequate one matches the one referred by the GOCCLES® glasses and the toluidine blue, only one biopsy will be made. Otherwise, two or three samples will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Rocío Teresa Martín Muñoz, Principal Investigator — Universidad Rey Juan Carlos de Madrid; Antonio Francisco López Sánchez, Study Director — Universidad Rey Juan Carlos de Madrid
Locations (1):
- Universidad Rey Juan Carlos de Madrid, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Scully C, Bagan J. Oral squamous cell carcinoma overview. Oral Oncol. 2009 Apr-May;45(4-5):301-8. doi: 10.1016/j.oraloncology.2009.01.004. Epub 2009 Feb 26. No abstract available. PMID 19249237
- [Background] Warnakulasuriya S. Causes of oral cancer--an appraisal of controversies. Br Dent J. 2009 Nov 28;207(10):471-5. doi: 10.1038/sj.bdj.2009.1009. PMID 19946320
- [Background] Warnakulasuriya S. Global epidemiology of oral and oropharyngeal cancer. Oral Oncol. 2009 Apr-May;45(4-5):309-16. doi: 10.1016/j.oraloncology.2008.06.002. Epub 2008 Sep 18. PMID 18804401
- [Background] McCullough MJ, Prasad G, Farah CS. Oral mucosal malignancy and potentially malignant lesions: an update on the epidemiology, risk factors, diagnosis and management. Aust Dent J. 2010 Jun;55 Suppl 1:61-5. doi: 10.1111/j.1834-7819.2010.01200.x. PMID 20553246
- [Background] Mignogna MD, Fedele S, Lo Russo L. The World Cancer Report and the burden of oral cancer. Eur J Cancer Prev. 2004 Apr;13(2):139-42. doi: 10.1097/00008469-200404000-00008. PMID 15100581
- [Background] Mello FW, Miguel AFP, Dutra KL, Porporatti AL, Warnakulasuriya S, Guerra ENS, Rivero ERC. Prevalence of oral potentially malignant disorders: A systematic review and meta-analysis. J Oral Pathol Med. 2018 Aug;47(7):633-640. doi: 10.1111/jop.12726. Epub 2018 Jun 6. PMID 29738071
- [Background] Warnakulasuriya S, Johnson NW, van der Waal I. Nomenclature and classification of potentially malignant disorders of the oral mucosa. J Oral Pathol Med. 2007 Nov;36(10):575-80. doi: 10.1111/j.1600-0714.2007.00582.x. PMID 17944749
- [Background] Farah CS, McIntosh L, Georgiou A, McCullough MJ. Efficacy of tissue autofluorescence imaging (VELScope) in the visualization of oral mucosal lesions. Head Neck. 2012 Jun;34(6):856-62. doi: 10.1002/hed.21834. Epub 2011 Aug 4. PMID 21818819
- [Background] Fedele S. Diagnostic aids in the screening of oral cancer. Head Neck Oncol. 2009 Jan 30;1:5. doi: 10.1186/1758-3284-1-5. PMID 19284694
- [Background] Scheer M, Neugebauer J, Derman A, Fuss J, Drebber U, Zoeller JE. Autofluorescence imaging of potentially malignant mucosa lesions. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2011 May;111(5):568-77. doi: 10.1016/j.tripleo.2010.12.010. Epub 2011 Mar 22. PMID 21429774
- [Background] Abati S, Bramati C, Bondi S, Lissoni A, Trimarchi M. Oral Cancer and Precancer: A Narrative Review on the Relevance of Early Diagnosis. Int J Environ Res Public Health. 2020 Dec 8;17(24):9160. doi: 10.3390/ijerph17249160. PMID 33302498
- [Background] Moro A, De Waure C, Di Nardo F, Spadari F, Mignogna MD, Giuliani M, Califano L, Gianni AB, Cardarelli L, Celentano A, Bombeccari G, Pelo S. The GOCCLES(R) medical device is effective in detecting oral cancer and dysplasia in dental clinical setting. Results from a multicentre clinical trial. Acta Otorhinolaryngol Ital. 2015 Dec;35(6):449-54. doi: 10.14639/0392-100X-922. PMID 26900252